CLINICAL TRIAL: NCT06645847
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Pilot Study to Evaluate the Effect of a Ketone Ester on Muscle and Immune Function in Older Men and Women Who Are at Risk for Strength and Mobility Decline
Brief Title: Targeting Aging With a Ketone Ester for Function in Frailty
Acronym: TAKEOFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buck Institute for Research on Aging (Other)
Collaborators: Ohio State University (Other); University of Connecticut (Other); California Pacific Medical Center Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024H0061
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Frail Elderly; Aging; Immune Function; Muscle Function
Keywords: ketone ester; exogenous ketone
MeSH Terms: interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Parallel group, randomized, double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study products will be allocated a code and labelled by an external team. The coding of the study products will be recorded and sealed in physical and electronic 'unblinding envelopes' that will only be opened by specific personnel if unblinding becomes necessary for subject safety. No one on the study team (including outcome assessor and statisticians) will be aware of the study product identity. The study products are matched for appearance, taste and calories and will not be visibly distinguishable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone ester (Active Comparator): Ketone ester (KE) (Chemical name: Bis-octanoyl-(R)-1,3-butanediol, Common name: C8 ketone di-ester) formulated as a dietary supplement.
  KE 12.5 g per day for 1 week; followed by KE 25 g per day for 1 week; followed by KE 37.5 g per day split into two doses for 1 week; followed by KE 50 g per day split into two doses for 17 weeks
  Interventions: Other: Ketone ester
- Non-ketone placebo (Placebo Comparator): Placebo oil (non-ketogenic canola oil) formulated as a dietary supplement. Placebo oil 12.5 g per day for 1 week; followed by Placebo oil 25 g per day for 1 week; followed by Placebo oil 37.5 g per day split into two doses for 1 week; followed by Placebo oil 50 g per day split into two doses for 17 weeks
  Interventions: Other: Placebo Comparator: Non-ketone placebo

INTERVENTIONS:
Other: Ketone ester — Ketone ester (KE) (Chemical name: Bis-octanoyl-(R)-1,3-butanediol, Common name: C8 ketone di-ester) formulated as a dietary supplement.
  KE 12.5 g per day for 1 week; followed by KE 25 g per day for 1 week; followed by KE 37.5 g per day split into two doses for 1 week; followed by KE 50 g per day split into two doses for 17 weeks
  Arms: Ketone ester
Other: Placebo Comparator: Non-ketone placebo — Placebo oil (non-ketogenic canola oil) formulated as a dietary supplement. Placebo oil 12.5 g per day for 1 week; followed by Placebo oil 25 g per day for 1 week; followed by Placebo oil 37.5 g per day split into two doses for 1 week; followed by Placebo oil 50 g per day split into two doses for 17 weeks
  Arms: Non-ketone placebo

SUMMARY:
This study aims to find out if a food supplement that contains a naturally occurring substance, ketones, can help to improve strength and general wellness in adults at, or over the age of 65 years who are experiencing a slight decline in their physical function.

Participation will involve a screening visit and 4 additional study visits over the course of 20 weeks. After being assessed for eligibility, study participants will be sorted into two groups at random and consume either a ketone or placebo supplement at home every day for 20 weeks. Both study products can cause gastro-intestinal side effects in some individuals. At all study visits, subjects will provide blood samples. At three study visits, subjects will be asked to complete physical performance tests, provide blood, stool and urine samples. They will also complete questionnaires during three study visits to assess physical function, markers of inflammation, and other aspects of general well-being.

The study enrolls at three sites across the United States, in California (Buck Institute), Ohio (Ohio State University), and Connecticut (University of Connecticut). The study is coordinated by the San Francisco Coordinating Center (California Pacific Medical Center).

DETAILED DESCRIPTION:
Screening (Phone and Visit 0):

Subjects are screened for eligibility by telephone for major exclusion criteria. They then attend a screening visit.

At the start of the visit subjects must meet pre-test requirements. During this visit, consent is obtained, followed by a medical history interview, a physical assessment and fasting blood samples are collected for screening analysis. Subjects who meet all the inclusion and none of the exclusion criteria will be scheduled for a Baseline (Visit 1) and at the end of Visit 1 will be randomized into one of the two experimental groups (ketone ester or placebo). Subjects will be shown and instructed on the use of the equipment for the physical function testing and complete a brief familiarization. A 24h diet log will be provided to complete before the next visit. A stool collection kit will also be provided along with use instructions to complete 3 days before Baseline visit.

Baseline Visit (Visit 1- Week 0):

Subjects must meet pre-test requirements. Changes to the subject's health and medication/supplement use will be assessed, and subject's compliance with inclusion/exclusion criteria will be reviewed. Fasted blood samples are collected. A clean catch urine sample is collected for archiving and additional plasma is banked for future aging biomarker analysis. After this a physical assessment will be conducted, including vital signs (after 5 minutes of rest), body weight and waist circumference. Investigators will reassess Katz's Activities of Daily Living (ADL) and Lawton's Instrumental Activities of Daily Living (IADLs) and CSHA Frailty Score (Canadian Study of Health and Aging). Then subjects will complete the following paper questionnaires: Profile of Mood States (Short form), Short Form Health Survey-36, Pittsburgh Sleep Quality Index, Pittsburgh Fatiguability Scale, Geriatric Depression Scale, Lower Urinary Tract Symptom Questionnaire. Subjects will complete cognitive function testing: Montreal Cognitive Assessment, Digit Symbol Substitution Task and Trails A and B. Subjects will complete physical function testing: Short Physical Performance Battery, 1 rep max leg press, sub maximal leg press repetitions to failure, 6-minute walk test and grip strength. Subjects will be given a stool sample collection kit to take home for at-home sample between Week 0 and 1; samples are returned by mail. Subject will be given a month's supply of study product to take home. Subjects will be reminded of study instructions (for study product consumption, daily Study Log completion, and to maintain habitual exercise, meal/diet, and medication/supplementation use). Subjects will be given a wearable actigraphy device and instructed on its use during the study.

At home procedures (Week 0 - 20):

Each day at home, subjects should consume their first meal of the day at a similar time and consume the study product with that first meal. For the first 7 days of the study, subjects will consume a 12.5 gram dose of study product. From day 8 onwards subjects will consume 25 grams of study product. From Week 3 onwards, they will consume a second serving (Week 3 = 12.5 grams, Week 4 - 20 = 25 grams) with their final meal of the day. The goal is to consume a 25 gram dose twice a day, one dose each with the first and last meal of the day. Subjects will complete the Study Log to confirm they consumed their study product. The Study Log will query the presence of specific symptoms in the hours after consumption of the study product with a beverage tolerance questionnaire (BTQ). Between days 6 - 9, subjects will collect a stool sample using the provided kit.

Every 2 weeks (excepting the site visits) the subjects will schedule a phone call with the Study Team in which they will verbally complete the BTQ for symptoms occurring in the preceding 2-week period. Compliance will be assessed, and AEs will also be assessed with an open-ended question. Subjects will be reminded of study instructions (for study product consumption, daily Study Log completion, and to maintain habitual exercise, meal/diet, and medication/supplementation use). After Week 16 check in, subjects will be mailed a stool sample collection kit for sample collection up to 3 days ahead of Visit 4.

From Week 5 onwards, a full BTQ is not completed daily. There is space in the Study Log to note any symptoms, these notes will be used to assess tolerance by interview for the previous 2-week interval; at Visit 2, during phone check-ins (Week 2, 6, 8, 10, 14, 16 and 18) and at Visits 3 and 4. Study product will be provided at one month intervals, it will be distributed directly during Visit 2 (week 4) and Visit 3 (week 12) and it will be shipped to subject's homes to arrive in week 8 and 16.

Intermediate Visit (Visit 2- Week 4): Subjects must meet pre-test requirements on arrival for Visit 2 (fasting ≥ 10 h, no alcohol ≥ 10 h, no exercise ≥ 10 h, no cannabis products ≥ 10 h); a reminder email (or telephone call if preferred by the subject) will be sent out ahead of the visit. On arrival, changes to medication/supplement use will be assessed, and the subject's compliance with inclusion/exclusion criteria will be reviewed. Subjects will be queried to ensure compliance with study instructions. Subjects will be asked to provide any unused product to assess compliance of Study Product consumption, and the Study Log (Part I) will be reviewed and collected. Adherence will be assessed, and adverse events (AEs) will also be assessed with an open-ended question. After this a physical assessment will be conducted, including vital signs (after 5 minutes of rest), body weight, body composition (using bioelectrical impedance), and waist circumference. Fasting blood samples will be collected for the following analysis: clinical chemistry, lipid panel, hematology and liver function. Additional samples will be retained to bank for possible future mechanistic investigations. Then, subjects will be asked to collect a urine sample for archiving. Subjects will verbally complete the BTQ for symptoms occurring in the preceding 2-week period.

Subjects will be reminded of study instructions (for study product consumption, daily Study Log completion, and to maintain habitual exercise, meal/diet, and medication/supplementation use). Subjects will be given a stool sample collection kit (instructions insert shown in Appendix) to take home for at-home sample collection up to 3 days after Visit 2, the stool sample will be returned to investigators using a prepaid mailer. Finally, subjects will be given a 4-week supply of study product to take home and Study Log (Part II). On this day, subjects will be asked to consume study products with their next meal after the test visit is complete.

Visit 3: Interim Endpoints Visit (Visit 4 - Week 12) and Final Visit (Visit 5- Week 20):

Follows identical testing procedures to Baseline Visit (Visit 3- Week 0).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 65 years of age, inclusive at Screening.
2. Passes the gait speed criteria at Screening.
3. Minimum body weight of 50 kgs at Screening.
4. Subject is willing and able to comply with all study procedures including randomization into any of the experimental groups, maintenance of habitual dietary intake, exercise and medication and supplement use, blood draws and the following prior to test visits: fasting (≥10 h; water only), no alcohol (≥ 10 h), no cannabis products (≥10 h) and no exercise (≥ 10 h).
5. Subject understands the study procedures and can provide informed consent to participate in the study.

Exclusion Criteria:

1. Subject is non ambulatory.
2. Subject has a CSHA clinical frailty score > 5.
3. Subject requires assistance with any activity of daily living, excluding continence.
4. Subject lives in an institutional setting (skilled nursing facility or residential care facility for the elderly).
5. Subject is a female who has not passed menopause.
6. Subject is unable to converse in English (or Spanish, if available at the study site).
7. Subject has been hospitalized within 30 days of Screening.
8. Subject has any physical limitation that would prevent them from performing 1RM leg press based on Medical Officer judgement.
9. Subject has an abnormal laboratory test result(s) of clinical importance at Screening, indicating unstable chronic disease of major organ dysfunction that requires urgent evaluation, at the discretion of the Medical Officer. One re-test will be allowed on a separate day prior to Visit 1, for subjects with abnormal laboratory test results. Additional clinical information may be gathered from the participant if needed to interpret the urgency of laboratory abnormalities (e.g. recent laboratory trends if an electrolyte is abnormal).
10. Subject has uncontrolled hypercholesterolemia on screening labs.
11. Subject has a history or presence of acute or uncontrolled and/or clinically active pulmonary (chronic obstructive pulmonary disease >= Gold 3), cardiac (e.g. >= New York Heart Association class III), hepatic (cirrhosis), renal (chronic kidney disease stage >= IIIb), endocrine (including type 1 diabetes), hematologic, immunologic, neurologic (e.g., Alzheimer's or Parkinson's diseases), psychiatric (including unstable depression and/or anxiety disorders) or biliary disorders. "Uncontrolled" and "clinically active" are per the judgement of the Medical Officer. Stable chronic disease is not an exclusion criterion unless specified. Chronic disease that is managed with the patient's physician per shared decision-making, even if sub optimally by typically recommended care, is not an exclusion criterion unless uncontrolled or clinically active.
12. Subject has a clinically important gastrointestinal condition that would potentially interfere with the evaluation of the study beverage [e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation, severe constipation (in the opinion of the Medical Officer), history of frequent diarrhea, history of surgery for weight loss, gastroparesis, systemic disease that might affect gut motility according to the Investigator, history of gastrointestinal ulcers or bleeding, history of pancreatitis, history of hiatal hernia, history of Barrett's esophagus, or history of esophageal cancer].
13. Heavy drinking (For women, 8 or more drinks per week. For men, 15 or more drinks per week).
14. Subject has a history of alcohol or substance abuse.
15. Subject has been instructed not to consume alcohol for medical reasons.
16. Subject has a known, clinically important allergy, intolerance, or sensitivity to any of the ingredients in the study beverages, including soy and milk protein.
17. Subject has uncontrolled hypertension as defined by the blood pressure measured at Screening. For subjects with elevated blood pressure at Screening, they are allowed for the purpose of this criteria to submit home readings from three separate days, or to have a repeat reading taken at the study site on a separate day before Visit 1.
18. Subject is undergoing treatment or active surveillance for cancer or has been diagnosed with cancer in the prior two years, except for non-melanoma skin cancer. Active surveillance is defined as regular imaging or laboratory tests at a frequency greater than annually. Cancer under long-term monitoring such as stable chronic lymphocytic leukemia need not be an exclusion, on the discretion of the Medical Officer.
19. Immunosuppressive disorders, taking immunosuppressive medications (including oral prednisone >10mg/day and biological immunosuppressants), or receiving chemotherapy.
20. Chronic antibiotic use (e.g. expected to be ongoing, regardless of frequency, throughout the study period).
21. Subject has extreme dietary habits (e.g., intermittent fasting or time restricted eating, Atkins diet, vegan, very high protein/low carbohydrate or has used weight-loss medications (including over-the-counter medications and/or supplements) or programs within 30 days of Screening.
22. Subject has followed a ketogenic diet or used ketone supplements (ketone salts or esters, and medium chain triglycerides) within 30 days of Screening.
23. Subject has a condition the Medical Officer believes would interfere with their ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.
24. Subject works nights or shifts that means it is not possible to maintain a consistent meal schedule during the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Frailty composite score | Baseline, 12 weeks, 20 weeks
  The primary outcome measure is the difference in the change in a four-item composite score of vigor-frailty (6 minute walk, 1 rep max leg press, digit symbol substitution, Pittsburg Fatigability Scale - Physical sub scale) over 20 weeks between groups. The original composite score was developed by the Study of Muscle Mass and Aging Group, it is continuous, and a higher score corresponds to better function.

SECONDARY OUTCOMES:
Tolerability key symptom index | 20 weeks
  Proportion of subjects reporting the same moderate to severe symptom (among dizziness, headache or nausea) occurring on more than one day within any given recall period (after week 0 - 2 acclimation period) when ketone esters are consumed daily for 20 weeks.
Safety Lab Tests | Baseline, Week 4, Week 12, 20 weeks
  Changes in clinical laboratory measurements when ketone esters are consumed daily for 20 weeks.
Leg fatigue - leg press at sub maximal weight | 20 weeks
  Difference in change in number of repetitions completed on the leg press machine at a sub maximal weight (subject must complete as many repetitions as they can).
Short Physical Performance Battery | Baseline, Week 12, 20 weeks
  Difference in change in Short Physical Performance Battery score
Grip Strength | Baseline, Week 12, Week 20
  Difference in change in grip strength measured by a hand grip dynamometer
Montreal Cognitive Assessment | Baseline, 12 weeks, 20 weeks
  Difference in change Montreal Cognitive Assessment score
Trails A and B | Baseline, Week 12, Week 20
  Standard trail making test scores between letters and numbers

OTHER OUTCOMES:
Immune phenotyping | 20 weeks
  Differences in cell subtypes, markers of immune aging and exhaustion, metabolite transporters and systemic inflammation.
Changes in gut microbial diversity | Baseline, Week 1, Week 4, Week 12, Week 20
  DNA sequencing of bacterial species in stool samples.
Profile of Mood States | Baseline, Week 12, Week 20
  Questionnaire about mood
Lower Urinary Tract Symptoms Questionnaire | Baseline, week 12, week 20
  Score on questionnaire assessing lower urinary tract symptoms
Short form 36 questionnaire | Baseline, Week 12, 20 weeks
  Quality of life questionnaire
Pittsburg Sleep Quality Index | Baseline, Week 12, Week 20
  Questionnaire about sleep quality
Geriatric Depression Scale | Baseline, Week 12, Week 20
  Questionnaire about mood
Skeletal muscle size (OSU only) | Baseline, 20 weeks
  Differences in muscle size measured by MRI
Skeletal muscle metabolites (OSU only) | Baseline, 20 weeks
  Differences in muscle metabolites measured by mass spectrometry
Resting metabolic rate (OSU only) | Baseline, Week 20
  Differences in resting metabolic rate measured by indirect calorimetry
Concentration of blood metabolites | Baseline, Week 4, Week 12
  Blood samples will be analyzed using targeted and un-targeted mass spectrometry to measure the concentration of metabolites that might be linked to aging. The difference in change over the study will be compared between groups.
Concentration of blood proteins | Baseline, Week 12, Week 20
  Blood samples will be analyzed using targeted and un-targeted mass spectrometry to measure the concentration of proteins that might be linked to aging. The difference in change over the study will be compared between groups.
Concentration of urine metabolites | Baseline, Week 12, week 20
  Urine samples will be analyzed using targeted and un-targeted mass spectrometry to measure the concentration of metabolites that might be linked to aging. The difference in change over the study will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: John Newman, MD, PhD, Principal Investigator — Buck Institute; Jeff Volek, Phd, Principal Investigator — Ohio State University; Jenna Bartley, PhD, Principal Investigator — University of Connecticut
Locations (3):
- United States (3):
  - Buck Institute for Research on Aging, Novato, California
  - UConn Health, Farmington, Connecticut
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stubbs BJ, Alvarez Azanedo G, Peralta S, Diaz SR, Gray W, Alexander L, Silverman-Martin W, Garcia TY, Blonquist TM, Upadhyay V, Turnbaugh PJ, Johnson JB, Newman JC. Rationale and protocol for a safety, tolerability and feasibility randomized, parallel arm, double-blind, placebo-controlled, pilot study of a novel ketone ester targeting frailty via immunometabolic geroscience mechanisms. PLoS One. 2024 Sep 18;19(9):e0307951. doi: 10.1371/journal.pone.0307951. eCollection 2024. PMID 39292659
- [Background] Crabtree CD, Blade T, Hyde PN, Buga A, Kackley ML, Sapper TN, Panda O, Roa-Diaz S, Anthony JC, Newman JC, Volek JS, Stubbs BJ. Bis Hexanoyl (R)-1,3-Butanediol, a Novel Ketogenic Ester, Acutely Increases Circulating r- and s-ss-Hydroxybutyrate Concentrations in Healthy Adults. J Am Nutr Assoc. 2023 Feb;42(2):169-177. doi: 10.1080/07315724.2021.2015476. Epub 2022 Mar 25. PMID 35512774
- [Background] Chen O, Blonquist TM, Mah E, Sanoshy K, Beckman D, Nieman KM, Winters BL, Anthony JC, Verdin E, Newman JC, Stubbs BJ. Tolerability and Safety of a Novel Ketogenic Ester, Bis-Hexanoyl (R)-1,3-Butanediol: A Randomized Controlled Trial in Healthy Adults. Nutrients. 2021 Jun 16;13(6):2066. doi: 10.3390/nu13062066. PMID 34208742